CLINICAL TRIAL: NCT06124157
Title: An International Pilot Study of Chemotherapy and Tyrosine Kinase Inhibitors With Blinatumomab in Patients With Newly-Diagnosed Philadelphia Chromosome-Positive or ABL-Class Philadelphia Chromosome-Like B-Cell Acute Lymphoblastic Leukemia
Brief Title: A Study Testing the Combination of Dasatinib or Imatinib to Chemotherapy Treatment With Blinatumomab for Children, Adolescents, and Young Adults With Philadelphia Chromosome Positive (Ph+) or ABL-Class Philadelphia Chromosome-Like (Ph-Like) B-cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-09214; NCI-2023-09214 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL2131 (Other: Children's Oncology Group); AALL2131 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2023-11-08; First posted 2023-11-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; Dasatinib; Daunorubicin; Doxorubicin; Imatinib Mesylate; Leucovorin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisolone; Methylprednisolone; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stratum I (Ph+ ALL) (Experimental): See detailed description
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Daunorubicin; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Drug: Vincristine
- Stratum II (PDGFRB ABL-Class fusions) (Experimental): See detailed description.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Imatinib; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine
- Stratum III (non-PDGFRB ABL-Class fusions) (Experimental): See detailed description.
  Interventions: Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Daunorubicin; Drug: Doxorubicin; Procedure: Echocardiography Test; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Drug: Pegaspargase; Drug: Prednisolone; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Receive IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Calaspargase Pegol — Receive IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
Drug: Cyclophosphamide — Receive IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Receive IV or subcutaneously
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Receive PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Stratum I (Ph+ ALL); Stratum III (non-PDGFRB ABL-Class fusions)
Drug: Daunorubicin — Receive IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Doxorubicin — Receive IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Imatinib — Given PO
  Arms: Stratum II (PDGFRB ABL-Class fusions)
Drug: Leucovorin — Receive PO or IV
  Other Names: Folinic acid
Drug: Mercaptopurine — Receive PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Receive IT or IV or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pegaspargase — Receive IV or intramuscularly
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisolone — Receive PO
  Other Names: (11beta)-11,17,21-Trihydroxypregna-1,4-diene-3,20-dione; .delta.1-Hydrocortisone; Adnisolone; Aprednislon; Capsoid; Cortalone; Cortisolone; Dacortin H; Decaprednil; Decortin H; Delta(1)Hydrocortisone; Delta- Cortef; Delta-Cortef; Delta-Diona; Delta-F; Delta-Phoricol; Delta1-dehydro-hydrocortisone; Deltacortril; Deltahydrocortisone; Deltasolone; Deltidrosol; Dhasolone; Di-Adreson-F; Dontisolon D; Estilsona; Fisopred; Frisolona; Gupisone; Hostacortin H; Hydeltra; Hydeltrasol; Klismacort; Kuhlprednon; Lenisolone; Lepi-Cortinolo; Linola-H N; Linola-H-Fett N; Longiprednil; Metacortandralone; Meti Derm; Meticortelone; Opredsone; Panafcortelone; Precortisyl; Pred-Clysma; Predeltilone; Predni-Coelin; Predni-Helvacort; Prednicortelone; Prednisolonum; Prelone; Prenilone; Sterane
Drug: Prednisone — Receive PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Stratum II (PDGFRB ABL-Class fusions); Stratum III (non-PDGFRB ABL-Class fusions)
Drug: Thioguanine — Receive PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
  Arms: Stratum II (PDGFRB ABL-Class fusions); Stratum III (non-PDGFRB ABL-Class fusions)
Drug: Vincristine — Receive IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine

SUMMARY:
This pilot trial assesses the effect of the combination of blinatumomab with dasatinib or imatinib and standard chemotherapy for treating patients with Philadelphia chromosome positive (Ph+) or ABL-class Philadelphia chromosome-like (Ph-like) B-Cell acute lymphoblastic leukemia (B-ALL). Blinatumomab is a bispecific antibody that binds to two different proteins-one on the surface of cancer cells and one on the surface of cells in the immune system. An antibody is a protein made by the immune system to help fight infections and other harmful processes/cells/molecules. Blinatumomab may bind to the cancer cell and a T cell (which plays a key role in the immune system's fighting response) at the same time. Blinatumomab may strengthen the immune system's ability to fight cancer cells by activating the body's own immune cells to destroy the tumor. Dasatinib and imatinib are in a class of medications called tyrosine kinase inhibitors. They work by blocking the action of an abnormal protein that signals cancer cells to multiply, which may help keep cancer cells from growing. Giving blinatumomab and dasatinib or imatinib in combination with standard chemotherapy may work better in treating patients with Ph+ or Ph-like ABL-class B-ALL than dasatinib or imatinib with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 3-year event free survival (EFS) of children, adolescents, and young adults <25 years old with newly-diagnosed Ph+ (BCR::ABL1-rearranged) B- ALL who are treated with a modified Berlin-Frankfurt-Münster (mBFM) chemotherapy backbone that incorporates three cycles of blinatumomab without traditional consolidation chemotherapy in combination with continuous dasatinib.

II. To estimate the 3-year EFS of children, adolescents, and young adults <25 years old with newly-diagnosed ABL-class Ph-like B-ALL who are treated with a modified BFM chemotherapy backbone that incorporates three cycles of blinatumomab without traditional consolidation chemotherapy in combination with continuous imatinib for those with PDGFRB gene fusions or dasatinib for those without PDGFRB gene fusions.

III. To describe the safety and toxicity profile (infections, mucositis, neurotoxicity, cytokine release syndrome, hypogammaglobulinemia, therapy delays > 14 days, and treatment-related mortality) for patients with Ph+ or ABL-class Ph-like B-ALL treated on this novel chemo-immunotherapy backbone with continuous tyrosine kinase inhibitor (TKI).

SECONDARY OBJECTIVES:

I. To estimate the 3-year overall survival (OS) of patients with Ph+ and ABL-class Ph-like B-ALL, respectively.

II. To estimate the 3-year EFS, disease-free survival (DFS), cumulative incidence rates (CIR) of relapse, and treatment related mortality (TRM), and OS of patients with ABL-class Ph-like B-ALL stratified by their underlying ABL-class fusion subtypes.

III. To describe rates of end of consolidation (EOC)/timepoint 2 (TP2) minimal residual disease (MRD) negativity defined as <1x10-4 or <0.01% for patients with Ph+ B-ALL.

IV. To describe rates of EOC/TP2 MRD negativity defined as <1x10-4 or <0.01% for patients with ABL-class Ph-like B-ALL collectively and based on their ABL-class fusion subtypes.

EXPLORATORY OBJECTIVES:

I. To describe rates of end of induction (EOI)/timepoint 1 (TP1) bone marrow MRD negativity defined as <1x10-4 or <0.01% with the introduction of the relevant TKI during Induction for patients with Ph+ and ABL-class Ph-like B-ALL, respectively.

II. To describe the outcomes of patients with Ph+ and ABL-class Ph-like B-ALL who are removed from protocol therapy due to Consolidation Failure.

III. To describe the percentage of patients with Ph+ and ABL-class Ph-like B-ALL who continue TKI beyond protocol-prescribed therapy and their outcomes.

IV. To describe the impact of MRD by next-generation sequencing (NGS) at End of Consolidation on outcomes for patients with Ph+ and ABL-class Ph-like B-ALL.

V. To describe the clinical characteristics and outcomes of patients with chronic myeloid leukemia-like biology.

VI. To describe the immune function of patients with Ph+ and ABL-class Ph-like B-ALL pre- and post-blinatumomab plus TKI and correlate with treatment response.

VII. To describe the TKI levels in the plasma and cerebrospinal fluid of children with Ph+ and ABL-class Ph-like B-ALL over the treatment course and correlate with outcome VIII. To describe the impact of TKIs and high-dose methotrexate interaction and identify clinical and biologic factors influencing methotrexate clearance.

OUTLINE:

STRATUM I (PH+ B-ALL PATIENTS):

INDUCTION PART I: Patients receive induction chemotherapy on days 1-14 as per standard of care (SOC).

INDUCTION PART II: Patients receive dasatinib PO once daily (QD) on days 15-29, daunorubicin intravenously (IV) over 15 minutes on days 15 and 22, prednisolone or prednisone PO twice daily (BID) on days 15-28, vincristine IV on days 15 and 22, methotrexate intrathecally (IT) on days 15, 22, and 29, and cytarabine IT on days 18 and 25 if central nervous system (CNS)-3 at study entry.

BLINATUMOMAB BLOCK I: Patients receive dexamethasone PO or intravenously (IV) on day 1, blinatumomab IV on days 1-28, dasatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study. Patients may undergo radiation therapy in 12 QD fractions.

BLINATUMOMAB BLOCK II: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV on days 1-28, dasatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study.

INTERIM MAINTENANCE I: Patients receive dasatinib PO QD until the end of interim maintenance I, mercaptopurine PO QD on days 1-56, vincristine IV on days 8, 22, 36, and 50, methotrexate IT on days 8 and 36, high-dose methotrexate IV over 24 hours on days 8, 22, 36 and 50, and leucovorin PO or IV on days 10, 11, 24, 25, 38, 39, 52 and 53 over 9 weeks on study.

BLINATUMOMAB BLOCK III: Patients receive blinatumomab IV on days 1-28, dasatinib PO QD on days 1-35, and methotrexate IT on day 1 over 5 weeks on study.

DELAYED INTENSIFICATION PART I: Patients receive dasatinib PO QD on days 1-28, methotrexate IT on day 1, dexamethasone PO or IV on days 1-7 and 15-21, doxorubicin IV over 15 minutes on days 1, 8, and 15, vincristine IV on days 1, 8, and 15, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on day 4 over 4 weeks on study.

DELAYED INTENSIFICATION PART II: Patients receive dasatinib PO QD on day 29 until the end of delayed intensification part II, cyclophosphamide IV over 60 minutes on day 29, cytarabine IV over 30 minutes on days 29-32 and 36-39, methotrexate IT on days 29 and 36, thioguanine PO on days 29-42, pegaspargase IV or calaspargase pegol on day 43 and vincristine IV on days 43 and 50 over 5 weeks on study.

INTERIM MAINTENANCE PART II: Patients receive dasatinib PO QD on day 1 until the end of interim maintenance part II, methotrexate IV on days 1, 11, 21, 31, and 41, vincristine IV on 1, 11, 21, 31, and 41, methotrexate IT on days 1 and 31, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on days 2, 22 or 23 over 8 weeks on study.

MAINTENANCE CYCLES I-II: Patients receive dasatinib PO QD on days 1-84, methotrexate IT on days 1 and 29, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study.

MAINTENANCE CYCLES III AND SUBSEQUENT CYCLES: Patients receive dasatinib PO QD on days 1-84, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study. Cycles repeat every 12 weeks for 2 years from the start of Induction therapy in the absence of disease progression or unacceptable toxicity.

STRATUM II (PDGFRB ABL-CLASS FUSIONS):

BLINATUMOMAB BLOCK I: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV on days 1-28, imatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study. Patients may undergo radiation therapy in 12 QD fractions.

BLINATUMOMAB BLOCK II: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV on days 1-28, imatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study.

INTERIM MAINTENANCE I: Patients receive imatinib PO QD until the end of interim maintenance I, mercaptopurine PO QD on days 1-56, vincristine IV on days 8, 22, 36, and 50, methotrexate IT on days 8 and 36, high-dose methotrexate IV over 24 hours on days 8, 22, 36 and 50, and leucovorin PO or IV on days 10, 11, 24, 25, 38, 39, 52 and 53 over 9 weeks on study.

BLINATUMOMAB BLOCK III: Patients receive blinatumomab IV on days 1-28, imatinib PO QD on days 1-35, and methotrexate IT on day 1 over 5 weeks on study.

DELAYED INTENSIFICATION PART I: Patients receive imatinib PO QD on days 1-28, methotrexate IT on day 1, dexamethasone PO or IV on days 1-7 and 15-21, doxorubicin IV over 15 minutes on days 1, 8, and 15, vincristine IV on days 1, 8, and 15, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on day 4 over 9 weeks on study.

DELAYED INTENSIFICATION PART II: Patients receive imatinib PO QD on day 29 until the end of Delayed Intensification part II, cyclophosphamide IV over 30-60 minutes on day 29, cytarabine IV over 30 minutes on days 29-32 and 36-39, methotrexate IT on days 29 and 36, thioguanine PO on days 29-42, and pegaspargase IV or calaspargase pegol IV on day 43, and vincristine IV on days 43 and 50 over 5 weeks on study.

INTERIM MAINTENANCE II: Patients receive imatinib PO QD until the end of interim maintenance II, methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, methotrexate IT on days 1 and 31, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on days 2, 22 or 23 over 8 weeks on study.

MAINTENANCE CYCLES I-II: Patients receive imatinib PO QD on days 1-84, methotrexate IT on days 1 and 29, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study.

MAINTENANCE CYCLES III AND SUBSEQUENT CYCLES: Patients receive imatinib PO QD on days 1-84, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study. Cycles repeat every 12 weeks for 2 years from the start of Induction therapy in the absence of disease progression or unacceptable toxicity.

STRATUM III (NON-PDGFRB ABL-CLASS FUSIONS):

BLINATUMOMAB BLOCK I: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV on days 1-28, dasatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study. Patients may undergo radiation therapy in 12 QD fractions.

BLINATUMOMAB BLOCK II: Patients receive dexamethasone PO or IV on day 1, blinatumomab IV on days 1-28, dasatinib PO on days 1-35, and methotrexate IT on days 1 and 15 over 5 weeks on study.

INTERIM MAINTENANCE I: Patients receive dasatinib PO QD until the end of interim maintenance I, mercaptopurine PO QD on days 1-56, vincristine IV on days 8, 22, 36, and 50, methotrexate IT on days 8 and 36, high-dose methotrexate IV over 24 hours on days 8, 22, 36 and 50, and leucovorin PO or IV on days 10, 11, 24, 25, 38, 39, 52 and 53 over 9 weeks on study.

BLINATUMOMAB BLOCK III: Patients receive blinatumomab IV on days 1-28, dasatinib PO on days 1-35, and methotrexate IT on day 1 over 5 weeks on study.

DELAYED INTENSIFICATION PART I: Patients receive dasatinib PO QD on days 1-28, methotrexate IT on day 1, dexamethasone PO or IV on days 1-7 and 15-21, doxorubicin IV over 15 minutes on days 1, 8, and 15, vincristine IV on days 1, 8, and 15, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on day 4 over 4 weeks on study.

DELAYED INTENSIFICATION PART II: Patients receive dasatinib PO QD and methotrexate IT on day 29 until the end of Delayed Intensification part II, cyclophosphamide IV over 30-60 minutes on day 29, cytarabine IV over 30 minutes on days 29-32 and 36-39, methotrexate IT on days 29 and 36, thioguanine PO on days 29-42, pegaspargase IV or calaspargase pegol on day 43 and vincristine IV on days 43 and 50 over 5 weeks on study.

INTERIM MAINTENANCE II: Patients receive dasatinib PO QD until the end of interim maintenance II, methotrexate IV and vincristine IV on days 1, 11, 21, 31 and 41, methotrexate IT on days 1 and 31, and pegaspargase IV or calaspargase pegol IV over 1-2 hours on days 2, 22 or 23 over 8 weeks on study.

MAINTENANCE CYCLES I-II: Patients receive dasatinib PO QD on days 1-84, methotrexate IT on days 1 and 29, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study.

MAINTENANCE CYCLES III AND SUBSEQUENT CYCLES: Patients receive dasatinib PO QD on days 1-84, methotrexate IT on day 1, dexamethasone PO BID or IV on days 1-5, 29-33, and 57-61, mercaptopurine PO on days 1-84, vincristine IV on days 1, 29 and 57, and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 on study. Cycles repeat every 12 weeks for 2 years from the start of Induction therapy in the absence of disease progression or unacceptable toxicity.

All patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening. Patients also undergo blood and cerebrospinal fluid (CSF) sample collection and bone marrow biopsy throughout the study and as clinically indicated on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 365 days and < 18 years (for AIEOP-BFM), > 365 days and < 22 years (for Children's Oncology Group [COG]) and > 365 days and < 46 years (for ALLTogether sites) at the time of enrollment
* Newly-diagnosed Ph+ or ABL-class Ph-like B-ALL. Leukemic blasts must express CD19. ABL-class fusions are defined as rearrangements involving the following genes predicted to be sensitive to imatinib and/or dasatinib: ABL1, ABL2, CSF1R, and PDGFRB
* Evidence of BCR::ABL1 should be documented by a clinically-validated assay prior to study entry on day 15 from the first dose of vinCRIStine during Induction therapy. ABL-class Ph-like B-ALL gene rearrangements should be documented by a clinically-validated assay and enrolled on study by day 1 of Blinatumomab Block 1. Accepted methods of detection include fluorescence in situ hybridization (FISH) using break-apart of colocalization signal probes, singleplex or multiplex reverse-transcription polymerase chain reaction (RT-PCR), whole-transcriptome or panel-based ribonucleic acid (RNA) sequencing (e.g., Hematologic Cancer Fusion Analysis, TruSight RNA Pan-Cancer Panel or equivalent). Confirmation of 5' fusion partner genes is not required for study enrollment
* Patients with Ph+ B-ALL must have previously started Induction therapy, which includes vinCRIStine, a corticosteroid, pegaspargase or calaspargase pegol, with or without anthracycline, and/or other standard cytotoxic chemotherapy
* Patients with Ph+ B-ALL have not received more than 14 days of systemic Induction therapy beginning with the first Induction dose of vinCRIStine
* Patients with ABL-class Ph-like B-ALL must have previously completed 4 or 5 weeks of multiagent Induction chemotherapy (Induction 1A)
* Patients may have started either imatinib or dasatinib prior to study entry but should have received no more than 14 days of TKI for Ph+ B-ALL or no more than 35 days of TKI for ABL-class Ph-like B-ALL
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of ≤ 2 or Karnofsky and Lansky performance scores ≥ 50%. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age
* For pediatric patients (age 1-17 years): a glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2, as determined by one of the following methods (must be performed within 7 days prior to enrollment unless otherwise indicated):

  * Estimated GFR (eGFR) ≥ 50 mL/min/1.73 m2
  * Measured GFR ≥ 50 mL/min/1.73 m^2 (any age). If measured GFR is used, it must be performed using direct measurement with a nuclear blood sampling method or small molecule clearance method (iothalamate or other molecule per institutional standard
* For adult patients (age 18 years or older): Creatinine clearance ≥ 30 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within 28 days prior to registration. Estimated creatinine clearance is based on body weight
* Direct bilirubin < 2.0 mg/dL (34.2 micromoles/L) (must be performed within 7 days prior to enrollment unless otherwise indicated)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 10 x upper limit of normal (ULN) (must be performed within 7 days prior to enrollment unless otherwise indicated)
* * Shortening fraction of ≥ 27% by echocardiogram (must be obtained within 21 days prior to enrollment and start of protocol therapy [repeat if necessary]) OR

  * Left Ventricular Ejection fraction of ≥ 50% by radionuclide angiogram or echocardiogram (must be obtained within 21 days prior to enrollment and start of protocol therapy [repeat if necessary]) AND
  * Corrected QT Interval, QTc < 480mSec (must be obtained within 21 days prior to enrollment and start of protocol therapy [repeat if necessary])

    * Note: Repeat echocardiogram and electrocardiogram are not required if they were performed at or after initial ALL diagnosis before study enrollment

Exclusion Criteria:

* Known history of chronic myeloid leukemia (CML)
* ABL-class Ph-like B-ALL who are CNS2 or CNS3 at end of Induction phase
* ALL developing after a previous cancer treated with cytotoxic chemotherapy
* Active, uncontrolled infection or active systemic illness that requires ongoing vasopressor support or mechanical ventilation
* Down syndrome (trisomy 21)
* Pregnancy and breast feeding

  * Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A negative pregnancy test is required for female patients of childbearing potential within 7 days prior to enrollment
  * Lactating females who plan to breastfeed their infants
  * Sexually active male and female patients of reproductive potential who have not agreed to use an effective contraception method for the duration of treatment according to protocol

    * NOTE: Patients who could become pregnant or could father a child must use effective contraception during protocol treatment and for 30 days after the last dose of dasatinib or 14 days after the last dose of imatinib dose or per institutional standard of care for multiagent chemotherapy, whichever is longer
* Prior treatment with TKIs before study entry with the exception of imatinib or dasatinib
* Patients with congenital long QT syndrome, history of ventricular arrhythmias, or heart block
* Patients with known Charcot-Marie-Tooth disease
* Patients with significant central nervous system pathology that would preclude treatment with blinatumomab, including history of severe neurologic disorder or autoimmune disease with central nervous system (CNS) involvement

  * Note: Patients with a history of seizures that are well controlled on stable doses of anti-epileptic drugs are eligible. Patients with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible. Patients with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved
* HIV-infected patients are eligible if on effective anti-retroviral therapy that does not interact with planned study agents and with undetectable viral load within 6 months of treatment
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 366 Days to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Philadelphia chromosome-positive (Ph+) (BCR::ABL1-rearranged) 3-year event free survival (EFS) | Time from enrollment to first event, relapse, second malignancy, or death in complete remission, or last contact for those who are event-free, assessed up to 3 years
  Will be assessed in children, adolescents, and young adults <25 years old with newly-diagnosed Ph+ (BCR::ABL1-rearranged) B acute lymphoblastic leukemia (B-ALL) who are treated with a modified Berlin-Frankfurt-Münster (mBFM) chemotherapy backbone that incorporates three cycles of blinatumomab without traditional consolidation chemotherapy in combination with continuous dasatinib. Will be estimated using the Kaplan-Meier method with standard errors of Peto.
ABL-class Ph-like B-ALL 3-year event free survival (EFS) | Time from enrollment to first event, relapse, second malignancy, or death in complete remission, or last contact for those who are event-free, assessed up to 3 years
  Will be assessed in children, adolescents, and young adults <25 years old with newly-diagnosed ABL-class Ph-like B-ALL who are treated with a modified BFM chemotherapy backbone that incorporates three cycles of blinatumomab without traditional consolidation chemotherapy in combination with continuous imatinib for those with PDGFRB gene fusions or dasatinib for those without PDGFRB gene fusions. Will be estimated using the Kaplan-Meier method with standard errors of Peto.
Incidence of adverse events | Up to 3 years
  Will assess the safety and toxicity profile (infections, mucositis, neurotoxicity, cytokine release syndrome, hypogammaglobulinemia, therapy delays > 14 days, and treatment-related mortality) for patients with Ph+ or ABL-class Ph-like B-ALL treated on this novel chemo-immunotherapy backbone with continuous tyrosine kinase inhibitor (TKI). Will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.

SECONDARY OUTCOMES:
3-year overall survival (OS) | Time from enrollment to death from any cause or date of last contact for those who are alive, assessed up to 3 years
  Will be assessed in patients with Ph+ and ABL-class Ph-like B-ALL, respectively. Will be estimated using the Kaplan-Meier method with standard errors of Peto.
3-year EFS | Time from enrollment to first event, relapse, second malignancy, or death in complete remission, or last contact for those who are event-free, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method with standard errors of Peto.
3-year disease free survival | Time from end of consolidation/blinatumomab block 2 (TP2) for early responders to first event (relapse, second malignancy, or death in complete remission) or last contact for those who are event-free, assessed up to 3 years
  Will be estimated using the Kaplan-Meier method with standard errors of Peto.
Cumulative incidence rates of relapse | Up to 3 years
Treatment related mortality | Up to 3 years
OS of patients with ABL-class Ph-like B-ALL | Time from enrollment to death from any cause or date of last contact for those who are alive, assessed up to 3 years
  Will be stratified by their underlying ABL-class fusion subtypes.
Rates of end of Consolidation (EOC)/timepoint 2 (TP2) minimal residual disease (MRD) negativity for patients with Ph+ B-ALL | From EOC to TP2
  Defined as <1x10^-4 or <0.01% for patients with Ph+ B-ALL.
Rates of EOC/TP2 MRD negativity for patients with ABL-class Ph-like B-ALL collectively and based on their ABL-class fusion subtypes | From EOC to TP2
  Defined as <1x10^-4 or <0.01% for patients with ABL-class Ph-like B-ALL collectively and based on their ABL-class fusion subtypes.

OTHER OUTCOMES:
Rates of end of induction (EOI)/timepoint 1 (TP1) bone marrow MRD negativity with the introduction of dasatinib | From EOI to TP1
  Defined as <1x10-4 or <0.01% with the introduction of the relevant TKI during Induction for patients with Ph+ B-ALL.
Outcomes of patients with Ph+ and Ph-like ABL-class B-ALL who are removed from protocol therapy due to consolidation failure | Up to 3 years
  Will be collected and described. A secondary analysis will also be conducted, examining the EFS of patients in both arms of the randomization using conventional definition of consolidation failure (EOC/TP2 MRD ≥ 1%).
Percentage of patients with Ph+ and ABL-class Ph-like B-ALL who continue TKI beyond protocol-prescribed therapy and their outcomes | Up to 3 years
Prognostic significance of MRD by next-generation sequencing (NGS) at end of induction and end of consolidation | Up to 3 years
  Its association with outcomes will be explored.
Clinical characteristics and outcomes of patients with chronic myeloid leukemia-like biology | Up to 3 years
  Will be summarized using descriptive statistics.
Immune function of Ph+ and ABL-class Ph-like B-ALL patients | Up to 3 years
TKI levels in the plasma and cerebrospinal fluid of children with Ph+ and ABL-class Ph-like B-ALL | Up to 3 years
Impact of TKIs and high-dose methotrexate interaction and identify clinical and biologic factors influencing methotrexate clearance | Up to 3 years
  Will be assessed by summarizing frequencies observed of the same.

CONTACTS AND LOCATIONS:
Overall Officials: Thai Hoa Tran, Principal Investigator — Children's Oncology Group
Locations (128):
- United States (117):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (8):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- University Pediatric Hospital, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm